CLINICAL TRIAL: NCT02161159
Title: An Observational Study of BOTOX® for the Management of Urinary Incontinence in Patients With Idiopathic Overactive Bladder
Acronym: GRACE
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/NS/OAB/002
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Urinary Incontinence; Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients With Urinary Incontinence Due to iOAB: Patients with urinary incontinence due to iOAB treated with BOTOX® in accordance with physician standard practice.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — botulinum toxin Type A administered in accordance with physician standard practice.
  Other Names: BOTOX®; onabotulinumtoxinA

SUMMARY:
This study will evaluate real world pattern of use of BOTOX® in actual clinical practice in patients with idiopathic overactive bladder (iOAB) with urinary incontinence whose symptoms have not been adequately managed by oral anticholinergic therapy.

ELIGIBILITY:
Inclusion Criteria:

* No prior treatment with botulinum toxin Type A for treatment of iOAB

Exclusion Criteria:

* Treatment with any botulinum toxin Type A within 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Urinary Incontinence Due to iOAB
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients Who have Greatly Improved or Improved on the 4-Point Treatment Benefit Scale (TBS) | Baseline, Week 12
Change From Baseline in Number of Urinary Incontinence Episodes | Baseline, Week 12

SECONDARY OUTCOMES:
Time to Re-Injection of BOTOX® | 12 Months
Number of Nocturia Episodes | 12 Months
Usage of Incontinence Support Products | 12 Months
Percentage of Patients Who Have at Least a 50% Reduction in Urinary Incontinence and Urinary Urgency Incontinence | Baseline, 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (53):
- Germany (32):
  - David Brix, Bad Mergentheim
  - Urologie Turmschtraße, Berlin
  - Uwe-Carsten, Berlin
  - Albrecht Kastein, Berlin
  - ATURO, Berlin
  - MVZ Burgdorf, Burgdorf, Hanover
  - Ev.-Luth. Diakonissenanstalt Dresden, Dresden
  - Stefan Carl, Emmendingen
  - Zentrum für Urologie FFM, Frankfurt
  - Georg-August-Universität Göttingen, Göttingen
  - Universitätsklinikum Halle (Saale), Halle
  - Urologikum Hamburg, Hamburg
  - Urologische Praxis Volksdorf, Hamburg
  - Claudia Olszak-Warnat, Herne
  - Westpfalz-Klinikum Kaiserslautern, Kaiserslautern
  - Urologie Zentrum Kiel, Kiel
  - Joachim Weiß, Lampertheim
  - Uro- Vital-Zentrum, GP Hellmeier, Krause et al, Landshut
  - Tom Kempe, Leipzig
  - Institut Dr. Schulze, Markkleeberg
  - Elke Stagge, Mülheim
  - Universitätsklinikum Münster, Münster
  - Urologen am Stadtpark, Nuremberg
  - Urologicum Osnabrück, Osnabrück
  - Simone Maier, Reutlingen
  - Andres Melchior, Salzatal OT Schiepzig
  - Andreas Reinhard Wicht, Sangerhausen
  - Franz Hirschle, Singen
  - Wolfgang Theurer, Stuttgart
  - Benjamin Fischer, Tuttlingen
  - Dietmar Jung, Tuttlingen
  - Kontinenzzentrum Südwest, Villingen-Schwenningen
- Spain (9):
  - Hospital Universitario Burgos, Burgos
  - Hospital de Cabueñes, Gijón
  - Hospital Virgen de la Victoria, Málaga
  - Complejo Hospitalario Universitario Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital de Valme, Seville
- Sweden (5):
  - Urologimottagningen, Hallands Sjukhus Halmstad, Halmstad
  - Urologiska kliniken, Södersjukhuset AB, Stockholm
  - Karolinska Hospital, Stockholm
  - Kvinnokliniken, Danderyds Sjukhus AB, Stockholm
  - Kirurgkliniken, Västervik Sjukhus, Västervik/Kalmar
- United Kingdom (7):
  - Queen Elizabeth Hospital, Queen Elizabeth Medical Centre, Edgbaston, Birmingham
  - Southern General Hospital, Glasgow, Lanarkshire
  - Leeds Teaching Hospitals NHS Trust, St. James's University Hospital, Leeds, West Yorkshire
  - University College London Hospitals NHS foundation Trust, London
  - Imperial College Healthcare NHS Trust, The Bays, St Mary's Hospital, London
  - St Helens & Knowsley Teaching Hospitals NHS Trust, Whiston Hospital, Prescot, Merseyside
  - Salisbury NHS Foundation Trust, Salisbury District Hospital, Salisbury, Wiltshire

REFERENCES:
- [Derived] Farrelly E, Hamid R, Lorenzo-Gomez MF, Schulte-Baukloh H, Yu J, Patel A, Nelson M. One treatment with onabotulinumtoxinA relieves symptoms of overactive bladder in patients refractory to one or more oral medications. Neurourol Urodyn. 2023 Aug;42(6):1203-1213. doi: 10.1002/nau.25221. Epub 2023 Jun 1. PMID 37260130
- [Derived] Poster. Female Pelvic Med Reconstr Surg. 2020 Oct 1;26(10S Suppl 1):S89-S189. doi: 10.1097/SPV.0000000000000936. No abstract available. PMID 33955921
- [Derived] Short orals. Female Pelvic Med Reconstr Surg. 2020 Oct 1;26(10S Suppl 1):S21-S77. doi: 10.1097/SPV.0000000000000934. No abstract available. PMID 33955918
- [Derived] Hamid R, Lorenzo-Gomez MF, Schulte-Baukloh H, Boroujerdi A, Patel A, Farrelly E. OnabotulinumtoxinA is a well tolerated and effective treatment for refractory overactive bladder in real-world practice. Int Urogynecol J. 2021 Jan;32(1):65-74. doi: 10.1007/s00192-020-04423-0. Epub 2020 Jul 27. PMID 32719964